CLINICAL TRIAL: NCT01968304
Title: Prospective Evaluation of Iron Status in Cancer Patients Beginning Chemotherapy
Acronym: CANFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2012/18
Record Dates: First submitted 2013-10-01; First posted 2013-10-24 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2015-11

CONDITIONS: Cancer
Keywords: Iron Status, Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Iron status follow up (No Intervention)
  Interventions: Other: Iron status follow up

INTERVENTIONS:
Other: Iron status follow up

SUMMARY:
In cancerology, anemia is a frequently-found situation, with a prevalence ranging from 30% to 90%, according to the series, disease stages, primary tumor locations and age (Scotte, Launay-Vacher et al. 2012). Although very probably a major cause of anemia, iron deficiency (ID) has been seldom investigated in the field of cancer. Its prevalence and incidence have never been assessed in a prospective study. It is well-known that anemia in the cancer setting is a source of asthenia and deterioration of quality of life, and can even reduce the efficacy of anticancer treatments such as radiotherapy. Correcting anemia therefore constitutes a daily challenge. Before 2004-2005, a very large proportion of patients were treated with erythropoietin (EPO). However, prescriptions for EPO appear to have considerably declined since the warnings issued by various scientific societies and governments on account of the possible increase in death rates and a higher incidence of thromboembolic events, as reported in 8 studies published to date (NCCN 2012). Simultaneously, the transfusion rate augmented from 3.4% to 8.7% and the median hemoglobin level fell from 10.8 to 8.9 g/dL (Feinberg, Bruno et al. 2012). The use of injectable iron appears to have improved the correction of anemia by EPO, as reported in several concordant studies versus oral iron and placebo (Pedrazzoli, Rosti et al. 2009; Steensma, Sloan et al. 2011). However, no monotherapy study has been conducted to evaluate the impact of injectable iron, alone without EPO, for the correction of ID (with or without anemia) in cancer treatment. Consequently, there exists a wide variety of practices, with an injectable iron prescription rate which, a priori, does not match the number of patients with iron deficiency. There exist other iron-based parameters to characterize ID but these are not yet used routinely during chemotherapy and need to be validated in the cancer field.

These parameters include:

* An assay of reticulocyte hemoglobin content (rHC)
* An assay of soluble transferrin receptor (sTfR) Soluble transferrin receptors are mainly located on red blood line cells receiving iron delivered by transferrin.

In this study, we propose to make a prospective assessment of the iron status of cancer patients beginning chemotherapy. The aim is to determine the proportion of patients who might benefit from injectable iron treatment. All ID will be covered prospectively over a 2-year period.

DETAILED DESCRIPTION:
Predictable risks The study will involve no increased risk or additional discomfort. Blood samples used in the study will be taken at blood samplings scheduled by the hospital practice of the reference institution. Only small amounts of blood will be taken for this study and they will have no repercussion on the patient's general status.

Evaluation of the expected results Improved knowledge of ID epidemiology in patients receiving chemotherapy would enable more effective targeting of potential patients specifically requiring management by injectable iron.

Expected benefits

Through the medium of this study :

* We hope to optimize ID screening, increase our knowledge of ID characteristics and enhance patient management.
* Management of anemia in the cancer setting could thus be modified, i.e. via injectable iron treatment involving no EPO, the dangers of which (increase in the number of thromboembolic events, and even its potentially negative impact on survival) are being more and more fully documented.
* Patients included in this study will benefit from the detection of ID, which otherwise would not have been discovered.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 18 years of age.
2. Patients with a locally advanced or metastatic solid cancer (breast, colorectal, prostate, ENT, and lung) scheduled to receive first-line chemotherapy for metastatic disease or Patients with a lymphoma-type hematologic cancer scheduled for first-line chemotherapy
3. Patients who have read the information leaflet and have signed the informed consent.
4. Patients covered by national medical insurance.

Exclusion Criteria:

1. Patients currently undergoing chemotherapy
2. Patients with diagnosed ID
3. Patients having received oral iron or injectable iron treatment during the previous 3 months
4. Patients receiving EPO or transfused during the 3 months prior to inclusion.
5. Patients unable to give their consent.
6. Patients over 18 but under guardianship or public guardianship.
7. Vulnerable individuals as defined by article L1121-5 to -8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
ID, whether absolute or functional, shall be defined according to the recommendations contained in NCCN 2012 (NCCN - Practice Guidelines in Oncology - version 2.2012) | 2015, december
  Absolute ID: ferritinemia < 30 ng/ml and saturation coefficient of transferrin < 15%,
  -Functional ID: ferritinemia < 800 ng/ml and transferrin saturation coefficient < 20%.
  Prevalence shall be represented by the ratio of the number of subjects with ID at commencement of chemotherapy over the total number of subjects present in the population at the same time.

SECONDARY OUTCOMES:
Incidence of ID during chemotherapy treatment at W6-W8 and W12-W14 | December 2015
  Incidence represents the occurrence rate of ID during chemotherapy at W6-W8 and W12-W14 over the total number of subjects present in the population during the week in question.
  Attention will also be given to the overall rate of patients with ID (prevalent patient rates and incident patient rates)
Changes in iron status in cancer patients receiving chemotherapy during W12-W14 | 2015, december
  For incident patients, i.e. those developing ID during their monitoring period, the time of occurrence and the duration of ID expressed in weeks will be evaluated.
  For prevalent patients, i.e. those with ID at commencement of chemotherapy, the duration of ID expressed in weeks will be evaluated. Note that patients presenting ID at W12-W14 will be offered treatment according to the currently implemented recommendations (NCCN - Practice Guidelines in Oncology - version 2.2012).The iron status evaluation will be continued with an additional sample-taking after 6 weeks (W18-W20) or 6 weeks following establishment of treatment.
Determination of the proportion of patients likely to benefit from injectable iron treatment | 2015, december
  Judgment criterion : Patients with absolute or functional ID at W12-W14 will be held to be candidates for injectable iron treatment The proportion of patients likely to benefit from injectable iron treatment will be determined on the basis of the prevalence and incidence results expressed as a percentage of the overall population
Characterization of the different iron parameters (hepcidin, chrome and soluble transferrin receptors) in order to define ID in the cancer setting | 2015, december
  These three iron parameters will be measured in the event of the patient presenting an ID as defined according to the above-mentioned criteria:
  * Hepcidin level,
  * Assay of the reticulyte hemoglobin content (rHC),
  * Soluble transferrin receptors (sTfR) sTfR/Log10 ferritin ratio.
Determination of the proportion of patients classified according to 4 categories (Q1,Q2,Q3,Q4) using the graph proposed by Steinmetz to assist prescribers when prescribing EPO and/or injectable iron | 2015, december
Determination of cancer pathologies and/or treatments predictive of occurrence of ID | 2015, december
Determination of the existence of a correlation between response to chemotherapy treatment and the presence of ID | 2015, december
  the overall response considered will be that determined by the patient's attending physician. Also, all criteria, whether biological (markers), clinical and/or scanographic (RECIST criteria for solid tumors and Cheason criteria for lymphomas), will be recorded. The tumor status will be classified according to 4 distinct categories: responding / stability / progression / reduction of tumor markers.
  The data regarding response to chemotherapy treatment, evaluated at the latest at W12-W14 in accordance with the usual standard management, shall be gathered and correlated with the presence, or not, of ID

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme BARRIERE, md, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine LACASSAGNE, Nice, France

REFERENCES:
- See also: Related Info — http://www.centreantoinelacassagne.org/